CLINICAL TRIAL: NCT03809650
Title: A Prospective, Multicenter, Open-label, Single Arm, Phase III Study to Assess the Efficacy and Safety of Macitentan (ACT-064992) in Subjects With Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Brief Title: A Clinical Study to Find Out if Macitentan is Effective and Safe in Japanese Patients With Chronic Thromboembolic Pulmonary Hypertension (CTEPH).
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a change in the development strategy
Sponsor: Actelion (Industry)
Collaborators: EPS Corporation (Other); Imepro Inc. (Unknown); General Laboratory, BML, Inc. (Unknown); Mitsubishi Logistics Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055E301
Record Dates: First submitted 2019-01-10; First posted 2019-01-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-03

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension (CTEPH)
Keywords: CTEPH; chronic thromboembolic pulmonary hypertension; macitentan
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label treatment period (Experimental): oral administration of macitentan 10 mg once daily
  Interventions: Drug: macitentan 10 mg

INTERVENTIONS:
Drug: macitentan 10 mg — macitentan 10 mg, film-coated tablet, oral use
  Other Names: ACT-064992, Opsumit®

SUMMARY:
The endothelin receptor antagonist macitentan showed significant improvement compared with placebo in pulmonary vascular resistance (PVR) and 6-minute walking distance (6MWD) in inoperable CTEPH patients in the phase II MERIT-1 trial (AC-055E201, NCT02021292). However, in the MERIT-1 trial Japanese patients were not included. Therefore, in line with Japan's medical environment, this phase III study is to confirm the efficacy and safety of macitentan in Japanese CTEPH patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study obtained from the subject or legal representative a) prior to initiation of any study mandated procedure
* Japanese subjects who have been diagnosed as having CTEPH:

  1. Subjects who have not undergone balloon pulmonary angioplasty (BPA) and for whom the investigator determines not to implement pulmonary endarterectomy (PEA) at the time of the acquisition of informed consent due to the organized thrombosis localized in the peripheral regions, high risk (complications, old age, etc.) or for any other reasons.
  2. Subjects who have postoperative persistent or recurrent pulmonary hypertension (PH) after undergoing pulmonary endarterectomy (PEA) and/or BPA.
* PH subjects whose WHO FC is I to IV
* 6MWD measured during the screening period ranges from 150 m to 450 m
* Subjects who meet the following conditions according to the right heart catheterization (RHC) performed during the screening period or within 8 weeks before the acquisition of the informed consent:

  1. Resting mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg
  2. Pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg (if PAWP cannot be measured or the value of PAWP is not reliable, left ventricular end-diastolic pressure ≤ 13 mmHg)
  3. Resting PVR ≥ 400 dyn*sec/cm5
* Subjects treated with anti-coagulation agents, unfractionated heparin or low molecular weight heparin at least 90 days prior to RHC at baseline
* Women with childbearing potential with negative serum pregnancy test results and able to follow the appropriate contraceptive methods from the date of starting the study drug administration up to 30 days after the discontinuation or completion of the study drug administration. Fertile male subjects able to use condom during the same period.

Exclusion Criteria:

* BPA within 90 days prior to undergoing baseline RHC
* PEA within 180 days prior to undergoing baseline RHC
* Subjects with unstable pulmonary hemodynamics who have postoperative persistent or recurrent PH after undergoing PEA and/or BPA
* Recurrent thromboembolism undergoing treatment with oral anti-coagulation agents
* Symptomatic acute pulmonary embolism within 180 days prior to the start of study drug administration
* Known moderate-to-severe restrictive lung disease or obstructive lung disease or known significant chronic lung disease diagnosed by chest imaging (e.g., interstitial lung disease, emphysema)
* Acute myocardial infarction during Screening period
* Severe liver impairment.
* Systolic blood pressure (SBP) < 90 mmHg at screening.
* Any known factor or disease that may interfere with treatment compliance or full participation in the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Evaluate the ratio in pulmonary vascular resistance (PVR) at rest from baseline to Week 16 | From Baseline to Week 16
  The resistance in the artery carrying blood to the lungs is called PVR. The PVR is the resistance in the artery carrying blood to the lungs and that has to be overcome by the right ventricle in heart in order to let blood flow to the lungs occur. The ratio in PVR at rest indicates the efficacy of macitentan in patients with CTEPH. The ratio in PVR at rest is calculated as PVR at Week 16 divided by baseline PVR. The ratio in PVR at rest from baseline to Week 16 of administration of macitentan is evaluated in subjects with CTEPH who are not indicated for pulmonary endarterectomy (PEA) and/or subjects who have postoperative persistent or recurrent pulmonary hypertension (PH) after PEA and/or balloon pulmonary angioplasty (BPA).

SECONDARY OUTCOMES:
Change from baseline to Week 16 in PVR at rest | From baseline to Week 16
  The PVR at rest will be calculated to evaluate the change in PVR at rest from pre-dosing (baseline) to post-dosing (Week 16).
Change from baseline to Week 16 in pulmonary vascular resistance index (PVRI) at rest | From baseline to Week 16
  The indexed PVR (PVRI) at rest will be calculated to evaluate the change in PVRI at rest from pre-dosing (baseline) to post-dosing (Week 16).
Change from baseline to Week 24 in 6-minute walk distance (6MWD) | From baseline to Week 24
  The purpose of the 6-minute walk is to test exercise tolerance and capacity. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. This endpoint evaluates the change in 6MWD from pre-dosing (baseline) to post-dosing (Week 24).
Change from baseline to Week 24 in Borg dyspnea index | From baseline to Week 24
  The Borg dyspnea index rates the severity of dyspnea (difficult or labored breathing) on a scale from 0 ('Nothing at all') to 10 ('Very, very severe - maximal'). A decrease in the Borg dyspnea index indicates an improvement. This endpoint evaluates the change in the Borg dyspnea index assessed at the end of measuring the 6MWD from pre-dosing (baseline) to post-dosing (Week 24).
Change from baseline to Week 24 in WHO functional class (WHO FC) | From baseline to Week 24
  This endpoint evaluates the change of WHO functional class from pre-dosing (baseline) to post-dosing (Week 24). Class I: no symptoms with exercise or at rest. No limitation of activity. Class II: No symptoms at rest but slight limitation with ordinary activities causing symptoms (e.g. short of breath with climbing a flight of stairs, grocery shopping, or making the bed). Class III: may not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. Class IV: symptoms at rest (e.g. dyspnea and/or fatigue) and inability to carry out any physical activity without symptoms. Patients in class IV manifest signs of right heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshinari Yokoyama, PhD, Study Director — Actelion Japan
Locations (23):
- Japan (23):
  - Fukuoka University Nishijin Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kagoshima University Hospital, Kagoshima
  - Nara Medical University Hospital, Kashihara
  - Kokura Kinen Hospital, Kitakyushu
  - Kobe University Hospital, Kobe
  - Saitama Cardiovascular and Respiratory Center, Kumagaya
  - Kure Kyosai Hospital, Kure
  - Kurume University Hospital, Kurume
  - Toho University Ohashi Medical Center, Meguro-ku
  - IIUHW Mita Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Okayama Medical Center, Okayama
  - Sapporo Medical University Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Sasebo City General Hospital, Sasebo
  - Keio University Hospital, Shinjuku-ku
  - National Cerebral and Cardiovascular Center Hospital, Suita
  - Mie University Hospital, Tsu
  - University of Tsukuba Hospital, Tsukuba
  - Yamagata University Hospital, Yamagata
  - Yokohama City University Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- See also: A Prospective, Multicenter, Open-label, Single Arm, Phase III Study to Assess the Efficacy and Safety of Macitentan (ACT-064992) in Subjects With Chronic Thromboembolic Pulmonary Hypertension (CTEPH) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=AC-055E301&attachmentIdentifier=aa227840-255d-4f06-8064-e8ebb89a846a&fileName=AC-055E301_CSR_Synopsis.pdf&versionIdentifier=